CLINICAL TRIAL: NCT03283475
Title: Surgical Management of Thigh Lipodystrophy
Brief Title: Different Surgical Modalities for Thigh Lipodystrophy Including Liposuction,Thigh Lift and Liposuction Assisted Thigh Lift
Acronym: thigh lift
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Gamal, plastic surgery department, Assiut University Hospital, Assiut, Egypt, Assiut University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13111987
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Thigh Lipodystrophy

STUDY DESIGN:
Intervention Model Description: The sample will be divided into two groups:- - Control group which will include 60 adult individuals between 18 and 35 years old who have BMI between 19 and 25, not complaining of any thigh contour deformities or skin redundancy with no history of body weight fluctuations. This group will be divided into two subgroups, 30 males and 30 females.
  The following measurements will be recorded :- Weight, height, thigh length, hip circumference, maximum buttocks circumference, upper thigh, middle thigh and lower thigh circumferences.
  - Patient group which will include 40 patients suffering from thigh lipodystrophy and contour deformities who will undergo surgical intervention after their assessment.
  After assessment, one of the following techniques will be selected:-
  * Liposuction only.
  * thigh lift.
  * Liposuction assisted thigh lift.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): - Control group will include 60 adult individuals between 18 and 35 years old who have body mass index (BMI) between 19 and 25, not complaining of any thigh contour deformities or skin redundancy with no history of body weight fluctuations. This group will be divided into two subgroups, 30 males and 30 females.
  The following measurements will be recorded :- Weight, height, thigh length, hip circumference, maximum buttocks circumference, upper thigh, middle thigh and lower thigh circumferences.
- patient group (Active Comparator): - Patient group will include 30 patients suffering from thigh lipodystrophy and contour deformities who will undergo surgical intervention after their assessment.
  After assessment, one of the following techniques will be selected:-
  * Liposuction only.
  * thigh lift.
  * Liposuction assisted thigh lift.
  Interventions: Procedure: thigh lift

INTERVENTIONS:
Procedure: thigh lift — liposuction-assisted medial avulsion thighplasty enables technically refined contouring of the thigh and the possible preservation of the local microvasculature, which results in reduced complication rates
  Other Names: thigh liposuction; liposuction assisted thigh lift
  Arms: patient group

SUMMARY:
The sample will be divided into two groups:- - Control group which will include 60 adult individuals between 18 and 35 years old who have BMI between 19 and 25, not complaining of any thigh contour deformities or skin redundancy with no history of body weight fluctuations. This group will be divided into two subgroups, 30 males and 30 females.

The following measurements will be recorded :- Weight, height, thigh length, hip circumference, maximum buttocks circumference, upper thigh, middle thigh and lower thigh circumferences.

- Patient group which will include 40 patients suffering from thigh lipodystrophy and contour deformities who will undergo surgical intervention after their assessment.

After assessment, one of the following techniques will be selected:-

* Liposuction only.
* thigh lift.
* Liposuction assisted thigh lift.

DETAILED DESCRIPTION:
Preoperative assessment:- Patients will be assessed regarding skin redundancy, history of weight loss and site of lipodystrophy whether deformity is proximal, distal or diffuse.

The same measurements mentioned above will be recorded for the patient group before surgery.

Preoperative photographs in anteroposterior, lateral and oblique positions will be taken.

Informed consent will be signed by the patient before surgery illustrating possible risks and complications of the surgery.

Postoperative assessment:- The outcomes will be evaluated 3 months after surgery regarding patient satisfaction and achievement of symmetry.

Early complications will be assessed within one week after surgery including hematoma, seroma, surgical site infection and wound dehiscence.

Late complications will be assessed at 3 months follow up including asymmetry, conspicuous scar and lymphedema.

Postoperative measurements and photographs will be recorded and compared with preoperative ones.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between18 and 35 years for control group and more than 18 years for patient group .
2. Patients with BMI between 19 and 25 for control group and less than 35 for patient group.

Exclusion Criteria:

1. Individuals less than 18 years.
2. Patients undergoing bariatric surgery within a period of less than one year.
3. Patients with BMI more than 35.
4. Patients with systemic illness as cancer or mental disorders & hepatic patients (generally debilitating diseases) or any contraindication for anesthesia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-05-14 (Actual); Primary Completion 2018-10-22 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
regarding patient satisfaction and achievement of symmetry. | 3 months
  questionnaire will be performed for the patient group to estimate degree of patient satisfaction with assessment of postoperative symmetry

SECONDARY OUTCOMES:
complication rates of different surgical techniques | 1 week and 3 months
  Early complications will be assessed within one week after surgery including hematoma, seroma, surgical site infection and wound dehiscence.
  Late complications will be assessed at 3 months follow up including asymmetry, conspicuous scar and lymphedema.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabbabe SW. Plastic Surgery after Massive Weight Loss. Mo Med. 2016 May-Jun;113(3):202-6. PMID 27443046
- [Result] Schmidt M, Pollhammer MS, Januszyk M, Duscher D, Huemer GM. Concomitant Liposuction Reduces Complications of Vertical Medial Thigh Lift in Massive Weight Loss Patients. Plast Reconstr Surg. 2016 Jun;137(6):1748-1757. doi: 10.1097/PRS.0000000000002194. PMID 27219231